CLINICAL TRIAL: NCT05803226
Title: Slow Art Plus: Developing and Piloting a Single Session Art Gallery-based Intervention for Mental Health Promotion Via a Mixed Method Waitlist Randomized Control Trial (RCT)
Brief Title: Slow Art Plus: A Single Session Art Gallery-based Intervention for Mental Health Promotion
Acronym: SAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanyang Technological University (Other)
Collaborators: National Gallery Singapore (Unknown)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Associate Professor of Psychology, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04IDP001152C430
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Mental Health Wellness 1; Self Care; Compassion
Keywords: Slow Looking; Mindfulness; Self-Compassion

STUDY DESIGN:
Intervention Model Description: The Slow Art Plus programme will involve a full 90-minute engagement, one that is built upon the existing Slow Art programme with added layers of mindfulness and self-compassion practices, as well as a response art activity that fosters symbolic dialogue and an emotional aesthetic experience between participants and the selected art piece.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The first 10-minute of Slow Art Plus involves a brief psychoeducation on slow looking, mindfulness, and self-compassion practices. This is followed by a 10-minute participants self-introduction and sharing of one act of self-kindness; a 10-minute facilitator led mindfulness meditation on affectionate breathing to foster greater somatic and emotional clarity for slow-looking. This is followed by a set of 30-minute slow looking activity with 1 selected art-piece, including: (a) creating an Artwork Title with one sentence description, (b) imaging music that resonates with the viewers' emotional response to artwork, and (c) sketching a Response Art that facilitates a dialogue between the viewer and the art piece for perspective widening. A 10-minute dyadic sharing follows with a 5-minute large group sharing of joint collective experience. Artwork reveal and sharing of its self-care implications is offered. Finally, a closure self-compassion activity of Supportive Healing Touch.
  Interventions: Behavioral: Slow Art Plus
- Control (No Intervention): Wait-list Control Arm who will receive the Slow Art Plus after the Experimental Arm completes the Intervention.

INTERVENTIONS:
Behavioral: Slow Art Plus — Slow Art Plus involved a full 90-minute engagement, one that is built upon the existing Slow Art programme with added layers of mindfulness and self-compassion practices, as well as a response art activity that fosters symbolic dialogue and an emotional aesthetic experience between participants and the selected artwork.
  Arms: Intervention

SUMMARY:
Utilizing a Participatory Action Research (PAR) paradigm, this 12-month study will adopt a mixed method Waitlist Randomized Control Trial (RCT) with a built-in acceptability and feasibility study to test the efficacy of Slow Art Plus in reducing stress and empowering self-care among 200 participants.

DETAILED DESCRIPTION:
The specific objectives are in four-folds: 1) To develop a standardized 90-minute single-session Slow Art Plus programme that integrates: (a) slow looking; (b) mindfulness meditation; (c) self-compassion activities; (d) reflective-creative expressions; and (e) dyadic sharing, to form a holistic mental health promotion intervention; 2) To assess the effectiveness of Slow Art Plus for reducing participants' perceived stress (primary outcomes); 3) To assess the effectiveness of Slow Art Plus for enhancing participants' self-awareness, self-care capacity, psychological resilience, and quality of life (secondary outcomes); and 4) To assess the feasibility and acceptability of the standardized Slow Art Plus protocol for large scale implementation in Singapore and greater Asia.

ELIGIBILITY:
Inclusion Criteria:

- individuals who can communicate in English and provide informed consent.

Exclusion Criteria:

* individuals who are suffering from depression or other major mental illness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Pre-Intervention
  The PSS comprises 10-items rated on a 5-point Likert scale and clustered into 2 subscales of perceived helplessness (e.g., "In the past couple of days, how often have you felt nervous and stressed today"), and perceived self-efficacy (e.g., In the past couple of days, how often have you felt that things were going your way"). The PSS possesses strong internal validity, reliability, and cross-cultural applicability.
Perceived Stress Scale (PSS) | Immediate Post Intervention
  The PSS comprises 10-items rated on a 5-point Likert scale and clustered into 2 subscales of perceived helplessness (e.g., "In the past couple of days, how often have you felt nervous and stressed today"), and perceived self-efficacy (e.g., In the past couple of days, how often have you felt that things were going your way"). The PSS possesses strong internal validity, reliability, and cross-cultural applicability.
Perceived Stress Scale (PSS) | 1-Day Follow-UP
  The PSS comprises 10-items rated on a 5-point Likert scale and clustered into 2 subscales of perceived helplessness (e.g., "In the past couple of days, how often have you felt nervous and stressed today"), and perceived self-efficacy (e.g., In the past couple of days, how often have you felt that things were going your way"). The PSS possesses strong internal validity, reliability, and cross-cultural applicability.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire Short Form (SF-FFMQ) | Pre-Intervention
  The SF-FFMQ comprises 20 items clustered into 5 subscales: (i) observe, (ii) describe, (iii) act with awareness, (iv) non-judging of inner experience, and (v) non-reactivity to inner experience. Higher scores indicating higher mindfulness capacity.
Five Facet Mindfulness Questionnaire Short Form (SF-FFMQ) | Immediate Post Intervention
  The SF-FFMQ comprises 20 items clustered into 5 subscales: (i) observe, (ii) describe, (iii) act with awareness, (iv) non-judging of inner experience, and (v) non-reactivity to inner experience. Higher scores indicating higher mindfulness capacity.
Five Facet Mindfulness Questionnaire Short Form (SF-FFMQ) | 1-Day Follow-Up
  The SF-FFMQ comprises 20 items clustered into 5 subscales: (i) observe, (ii) describe, (iii) act with awareness, (iv) non-judging of inner experience, and (v) non-reactivity to inner experience. Higher scores indicating higher mindfulness capacity.
Self-Compassion Scale - Short Form (SCS-SF) | Pre-Intervention
  The SCS-SF comprises 12 items clustered into 6 subscales: (i) self-kindness, (ii) common humanity, (iii) mindfulness, (iv) self-judgement, (v) isolation, and (iv) over-identification. Higher scores indicating higher self-compassion capacity.
Self-Compassion Scale - Short Form (SCS-SF) | Immediate Post Intervention
  The SCS-SF comprises 12 items clustered into 6 subscales: (i) self-kindness, (ii) common humanity, (iii) mindfulness, (iv) self-judgement, (v) isolation, and (iv) over-identification. Higher scores indicating higher self-compassion capacity.
Self-Compassion Scale - Short Form (SCS-SF) | 1-Day Follow-Up
  The SCS-SF comprises 12 items clustered into 6 subscales: (i) self-kindness, (ii) common humanity, (iii) mindfulness, (iv) self-judgement, (v) isolation, and (iv) over-identification. Higher scores indicating higher self-compassion capacity.
Ego-Resilience Scale-11 (ER-11) | Pre-Intervention
  The ER-11 comprises 11-items clustered into 3 subscales: (i) active engagement with the world, (ii) repertoire of problem-solving strategies, and (iii) integrated performance under stress. Higher scores indicating higher ego-resilience.
Ego-Resilience Scale-11 (ER-11) | Immediate Post Intervention
  The ER-11 comprises 11-items clustered into 3 subscales: (i) active engagement with the world, (ii) repertoire of problem-solving strategies, and (iii) integrated performance under stress. Higher scores indicating higher ego-resilience.
Ego-Resilience Scale-11 (ER-11) | 1-Day Follow-Up
  The ER-11 comprises 11-items clustered into 3 subscales: (i) active engagement with the world, (ii) repertoire of problem-solving strategies, and (iii) integrated performance under stress. Higher scores indicating higher ego-resilience.
Single-Item Quality of Life Scale (SI-QOLS) | Pre-Intervention
  1 item measures quality of life. Higher scores indicating higher QOL.
Single-Item Quality of Life Scale (SI-QOLS) | Immediate Post Intervention
  1 item measures quality of life. Higher scores indicating higher QOL.
Single-Item Quality of Life Scale (SI-QOLS) | 1-Day Follow-Up
  1 item measures quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Andy HY Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho AHY, Ma SHX, Ng JT, Choo PY, Tan-Ho G, Pooh KCL, Teng A. Slow art plus: developing and piloting a single session art gallery-based intervention for mental health promotion via a mixed method waitlist randomized control trial. Front Public Health. 2024 May 13;12:1238564. doi: 10.3389/fpubh.2024.1238564. eCollection 2024. PMID 38803811